CLINICAL TRIAL: NCT05847751
Title: The Use of ACURATE Neo 2 Valve in Patients With Symptomatic Aortic Valve Stenosis
Acronym: BSC07
Status: Active, not recruiting | Type: Observational
Sponsor: Ceric Sàrl (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Other Study IDs: MENA TAVI
Record Dates: First submitted 2023-03-01; First posted 2023-05-08 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Severe Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Aortic valve replacement — Trans Aortic Valve Replacement (TAVI)

SUMMARY:
The objective of this study is to evaluate the ACURATE Neo2 in the Middle East population with severe, symptomatic aortic stenosis.

DETAILED DESCRIPTION:
The MENA-TAVI study is an investigator-initiated, prospective, single-arm observational trial.

Patients referred for or presenting with severe aortic stenosis requiring an intervention constitute the source population. The Heart Team consisting of interventional cardiologists and cardiovascular surgeons will evaluate the patients by integrating the available clinical data, the predicted 30-day mortality, individual factors affecting mortality such as frailty as well as the estimated life-expectancy and the patient's wishes to finally reach a consensus on the optimal treatment strategy with regards to transcatheter or surgical aortic valve replacement. Patients planned for TAVI will be screened for eligibility. If patients fulfill all inclusion and do not meet exclusion criteria, they will be informed about the study's purpose and course and will be asked for participation and written informed consent. In case of consent, they will be treated by the ACURATE neo2 aortic bioprosthesis.

At discharge and at 30 days, the clinical outcomes composing the primary safety endpoint will be captured. Additional clinical, procedural and echocardiographic data will be obtained at discharge and at 30 days for assessment of secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Subject will be included if all of the following criteria are met:

  * Patient with severe aortic stenosis defined by an aortic valve area (AVA) < 1cm2 or AVA indexed to body surface area (BSA) of < 0.6 cm2/m2, including low-flow severe aortic stenosis defined by stroke volume index (SVI) < 35ml/m2, as assessed by integration of echocardiographic and invasive measurements
  * Subject is symptomatic (heart failure symptoms with New York Heart Association (NYHA) Functional Class > I, angina or syncope)
  * Patient is considered at high (STS-PROM (Society of Thoracic Surgeons-Predicted Risk of Mortality) score >8) or intermediate (STS-PROM score >4) risk by the Heart Team.
  * The heart team agrees on eligibility of the patient for participation and that TAVR (Transcatheter aortic valve replacement) (TAVR) by transfemoral access constitutes the most appropriate treatment modality, from which the patient will likely benefit most
  * Aortic annulus dimensions suitable (area range: 338-573 mm2 AND perimeter range: 66-85 mm) based on ECG-gated multislice computed tomographic measurements. Findings of transesophageal echocardiography (TEE) and conventional aortography should be integrated in the anatomic assessment if available
  * Arterial aorto-iliac-femoral axis suitable for transfemoral access with a minimum access vessel diameter ≥ 6 mm as assessed by multislice computed tomographic angiography and/or conventional angiography
  * Written informed consent of the patient or her/his legal representative
  * Patient understands the purpose, the potential risks as well as benefits of the trial and is willing to participate in all parts of the follow-up

Exclusion Criteria:

* Subject will not be included if any one of the following conditions exists:

  * Non-valvular aortic stenosis
  * Congenital aortic stenosis or unicuspid or bicuspid aortic valve
  * Non-calcific acquired aortic stenosis
  * Anatomy not appropriate for transfemoral transcatheter aortic valve implantation due to size of the aortic annulus or degree or eccentricity of calcification of the native aortic valve or tortuosity of the aorta or ilio-femoral arteries
  * Emergency procedure including patients in cardiogenic shock (low cardiac output, vasopressor dependence, mechanical hemodynamic support)
  * Severely reduced left ventricular (LV) function (ejection fraction < 20%)
  * Pre-existing prosthetic heart valve in aortic position
  * Presence of mitral valve prosthesis
  * Concomitant planned procedure except for percutaneous coronary intervention (PCI)
  * Planned non-cardiac surgery within 30 days
  * Stroke within 30 days of the procedure.
  * Myocardial infarction within 30 days of the procedure (except type 2)
  * Evidence of intra-cardiac mass, thrombus or vegetation
  * Severe coagulation conditions
  * Inability to tolerate anticoagulation/anti-platelet therapy
  * Active bacterial endocarditis or other active infections
  * Hypertrophic cardiomyopathy
  * Contraindication to contrast media or allergy to nitinol
  * Participation in another trial, which would lead to deviations in the preparation or performance of the intervention or the post-implantation management from this protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 100 patients from Middle East population with severe, symptomatic aortic stenosis will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | Post-procedure discharge of patient from the hospital (Preferably 1- 3 days post procedure)
  All deaths reported
Any stroke (disabling and non-disabling) | Post-procedure discharge of patient from the hospital (Preferably 1- 3 days post procedure)
  All stroke events

SECONDARY OUTCOMES:
Technical success as defined by VARC-3 | Post-procedure discharge of patient from the hospital (Preferably 1- 3 days post procedure)
  Combined endpoint composed of:
  * Freedom from mortality
  * Successful access, delivery of the device, and retrieval of the delivery system
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location
  * Freedom from surgery or intervention related to the device or to a major vascular or access-related, or cardiac structural complication
Device success as defined by VARC-3 | Post-procedure discharge of patient from the hospital and at 30 days follow up
  Combined endpoint composed of:
  * Technical success
  * Freedom from mortality
  * Freedom from surgery or intervention related to the device or to a major vascular or access related or cardiac structural complication
  * Intended performance of the valve (mean gradient <20mmHg, peak velocity <3 m/s, Doppler velocity index ≥0.25, and less than moderate aortic regurgitation)
Early safety as defined by VARC-3 | At 30 days
  Combined endpoint composed of:
  * Freedom from all-cause mortality
  * Freedom from all stroke
  * Freedom from VARC 3 type 2-4 bleeding
  * Freedom from major vascular, access-related, or cardiac structural complication
  * Freedom from acute kidney injury stage 3 or 4
  * Freedom from moderate or severe aortic regurgitation
  * Freedom from new permanent pacemaker due to procedure related conduction abnormalities
  * Freedom from surgery or intervention related to the device
Modified combined early safety and clinical efficacy at 30 days as defined by the Valve Academic research Consortium (VARC-2) | At 30 days
  * All cause death)
  * All stroke (disabling and non-disabling)
  * Acute kidney injury (Stage 1 or 2, including renal replacement therapy)
  * Coronary artery obstruction requiring intervention
  * Major vascular complication
  * Valve related dysfunction requiring repeat procedure
  * Re-hospitalization for valve related symptoms or worsening congestive heart failure
  * Valve related dysfunction
  * Prosthetic aorta valve stenosis: mean aortic valve gradient >= 20 mmHg, effective orifice area (EOL) <= 1.1 cm2 (if body surface area >=1.6 m2) or <= 0.9 cm2 if BSA <1.6 m2 and/or Doppler velocity index <0.35
  * Moderate or severe prosthetic valve regurgitation according to VARC-2
Clinical efficacy as defined by VARC-3 | At 30 days
  Combined endpoint composed of:
  * Freedom from all-cause mortality
  * Freedom from all stroke
  * Freedom from hospitalization for procedure- or valve-related causes
  Combined endpoint composed of:
  * Freedom from all-cause mortality
  * Freedom from all stroke
  * Freedom from hospitalization for procedure- or valve-related causes
All-cause mortality | At 30 days
  All deaths reported
Valve-related mortality | At 30 days
  All deaths related to valve
All stroke (ischaemic, haemorrhagic) | At 30 days
  All stroke reported
Hospitalization (or re-hospitalization) | At 30 days
  All hospitalization reported
Bleeding and transfusions (VARC3 type 1 - 4) | At 30 days
  All bleeding events reported
Bioprosthetic valve dysfunction | At 30 days
  (structural, non structural, thrombosis, endocarditis): (Stage 1 to 3)
Clinically significant prosthetic valve thrombosis | At 30 days
  Valve related thrombosis
Implantation of permanent pacemaker | At 30 days
  Pacemaker implantation
Occurrence of atrial fibrilation | At 30 days
  atrial fbrillation reported

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed BALGHITH, MD, Principal Investigator — King Fahad National Guard Hospital
Locations (7):
- Egypt (3):
  - Magdy Yacoub heart center, Aswān
  - Ain shams Specialized hospital, Cairo
  - Badr hospital, Cairo
- American University of Beirut, Beirut, Lebanon
- Saudi Arabia (3):
  - King Fahad Armed Forces Hospital, Jeddah
  - King Fahad National Guard Hospital, Riyadh
  - National Guard Hospital - King Abdulaziz Medical City, Riyadh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iung B, Baron G, Butchart EG, Delahaye F, Gohlke-Barwolf C, Levang OW, Tornos P, Vanoverschelde JL, Vermeer F, Boersma E, Ravaud P, Vahanian A. A prospective survey of patients with valvular heart disease in Europe: The Euro Heart Survey on Valvular Heart Disease. Eur Heart J. 2003 Jul;24(13):1231-43. doi: 10.1016/s0195-668x(03)00201-x. PMID 12831818
- [Background] Otto CM, Prendergast B. Aortic-valve stenosis--from patients at risk to severe valve obstruction. N Engl J Med. 2014 Aug 21;371(8):744-56. doi: 10.1056/NEJMra1313875. No abstract available. PMID 25140960
- [Background] Tibazarwa KB, Volmink JA, Mayosi BM. Incidence of acute rheumatic fever in the world: a systematic review of population-based studies. Heart. 2008 Dec;94(12):1534-40. doi: 10.1136/hrt.2007.141309. Epub 2008 Jul 31. PMID 18669552
- [Background] Marijon E, Mirabel M, Celermajer DS, Jouven X. Rheumatic heart disease. Lancet. 2012 Mar 10;379(9819):953-964. doi: 10.1016/S0140-6736(11)61171-9. PMID 22405798
- [Background] Otto CM, Lind BK, Kitzman DW, Gersh BJ, Siscovick DS. Association of aortic-valve sclerosis with cardiovascular mortality and morbidity in the elderly. N Engl J Med. 1999 Jul 15;341(3):142-7. doi: 10.1056/NEJM199907153410302. PMID 10403851
- [Background] Otto CM. Calcific aortic stenosis--time to look more closely at the valve. N Engl J Med. 2008 Sep 25;359(13):1395-8. doi: 10.1056/NEJMe0807001. No abstract available. PMID 18815402
- [Background] Thanassoulis G, Campbell CY, Owens DS, Smith JG, Smith AV, Peloso GM, Kerr KF, Pechlivanis S, Budoff MJ, Harris TB, Malhotra R, O'Brien KD, Kamstrup PR, Nordestgaard BG, Tybjaerg-Hansen A, Allison MA, Aspelund T, Criqui MH, Heckbert SR, Hwang SJ, Liu Y, Sjogren M, van der Pals J, Kalsch H, Muhleisen TW, Nothen MM, Cupples LA, Caslake M, Di Angelantonio E, Danesh J, Rotter JI, Sigurdsson S, Wong Q, Erbel R, Kathiresan S, Melander O, Gudnason V, O'Donnell CJ, Post WS; CHARGE Extracoronary Calcium Working Group. Genetic associations with valvular calcification and aortic stenosis. N Engl J Med. 2013 Feb 7;368(6):503-12. doi: 10.1056/NEJMoa1109034. PMID 23388002
- [Background] Katz R, Wong ND, Kronmal R, Takasu J, Shavelle DM, Probstfield JL, Bertoni AG, Budoff MJ, O'Brien KD. Features of the metabolic syndrome and diabetes mellitus as predictors of aortic valve calcification in the Multi-Ethnic Study of Atherosclerosis. Circulation. 2006 May 2;113(17):2113-9. doi: 10.1161/CIRCULATIONAHA.105.598086. Epub 2006 Apr 24. PMID 16636166
- [Background] Owens DS, Katz R, Takasu J, Kronmal R, Budoff MJ, O'Brien KD. Incidence and progression of aortic valve calcium in the Multi-ethnic Study of Atherosclerosis (MESA). Am J Cardiol. 2010 Mar 1;105(5):701-8. doi: 10.1016/j.amjcard.2009.10.071. PMID 20185020
- [Background] Iung B, Vahanian A. Degenerative calcific aortic stenosis: a natural history. Heart. 2012 Nov;98 Suppl 4:iv7-13. doi: 10.1136/heartjnl-2012-302395. PMID 23143128
- [Background] Makkar RR, Fontana GP, Jilaihawi H, Kapadia S, Pichard AD, Douglas PS, Thourani VH, Babaliaros VC, Webb JG, Herrmann HC, Bavaria JE, Kodali S, Brown DL, Bowers B, Dewey TM, Svensson LG, Tuzcu M, Moses JW, Williams MR, Siegel RJ, Akin JJ, Anderson WN, Pocock S, Smith CR, Leon MB; PARTNER Trial Investigators. Transcatheter aortic-valve replacement for inoperable severe aortic stenosis. N Engl J Med. 2012 May 3;366(18):1696-704. doi: 10.1056/NEJMoa1202277. Epub 2012 Mar 26. PMID 22443478
- [Background] Rosenhek R, Zilberszac R, Schemper M, Czerny M, Mundigler G, Graf S, Bergler-Klein J, Grimm M, Gabriel H, Maurer G. Natural history of very severe aortic stenosis. Circulation. 2010 Jan 5;121(1):151-6. doi: 10.1161/CIRCULATIONAHA.109.894170. Epub 2009 Dec 21. PMID 20026771
- [Background] Clark MA, Arnold SV, Duhay FG, Thompson AK, Keyes MJ, Svensson LG, Bonow RO, Stockwell BT, Cohen DJ. Five-year clinical and economic outcomes among patients with medically managed severe aortic stenosis: results from a Medicare claims analysis. Circ Cardiovasc Qual Outcomes. 2012 Sep 1;5(5):697-704. doi: 10.1161/CIRCOUTCOMES.112.966002. Epub 2012 Sep 4. PMID 22949492
- [Background] Braunwald E. On the natural history of severe aortic stenosis. J Am Coll Cardiol. 1990 Apr;15(5):1018-20. doi: 10.1016/0735-1097(90)90235-h. No abstract available. PMID 2312955
- [Background] Teo KK, Corsi DJ, Tam JW, Dumesnil JG, Chan KL. Lipid lowering on progression of mild to moderate aortic stenosis: meta-analysis of the randomized placebo-controlled clinical trials on 2344 patients. Can J Cardiol. 2011 Nov-Dec;27(6):800-8. doi: 10.1016/j.cjca.2011.03.012. Epub 2011 Jul 13. PMID 21742465
- [Background] Rossebo AB, Pedersen TR, Boman K, Brudi P, Chambers JB, Egstrup K, Gerdts E, Gohlke-Barwolf C, Holme I, Kesaniemi YA, Malbecq W, Nienaber CA, Ray S, Skjaerpe T, Wachtell K, Willenheimer R; SEAS Investigators. Intensive lipid lowering with simvastatin and ezetimibe in aortic stenosis. N Engl J Med. 2008 Sep 25;359(13):1343-56. doi: 10.1056/NEJMoa0804602. Epub 2008 Sep 2. PMID 18765433
- [Background] Watkins DA, Johnson CO, Colquhoun SM, Karthikeyan G, Beaton A, Bukhman G, Forouzanfar MH, Longenecker CT, Mayosi BM, Mensah GA, Nascimento BR, Ribeiro ALP, Sable CA, Steer AC, Naghavi M, Mokdad AH, Murray CJL, Vos T, Carapetis JR, Roth GA. Global, Regional, and National Burden of Rheumatic Heart Disease, 1990-2015. N Engl J Med. 2017 Aug 24;377(8):713-722. doi: 10.1056/NEJMoa1603693. PMID 28834488
- [Background] Vahanian A, et al. The ESC Textbook of Cardiovascular Medicine. 2nd ed. Oxford: Oxford University Press; 2009, pp 625-70.
- [Background] Dewey TM, Brown D, Ryan WH, Herbert MA, Prince SL, Mack MJ. Reliability of risk algorithms in predicting early and late operative outcomes in high-risk patients undergoing aortic valve replacement. J Thorac Cardiovasc Surg. 2008 Jan;135(1):180-7. doi: 10.1016/j.jtcvs.2007.09.011. Epub 2007 Nov 26. PMID 18179938
- [Background] Brown JM, O'Brien SM, Wu C, Sikora JA, Griffith BP, Gammie JS. Isolated aortic valve replacement in North America comprising 108,687 patients in 10 years: changes in risks, valve types, and outcomes in the Society of Thoracic Surgeons National Database. J Thorac Cardiovasc Surg. 2009 Jan;137(1):82-90. doi: 10.1016/j.jtcvs.2008.08.015. PMID 19154908
- [Background] Chukwuemeka A, Borger MA, Ivanov J, Armstrong S, Feindel CM, David TE. Valve surgery in octogenarians: a safe option with good medium-term results. J Heart Valve Dis. 2006 Mar;15(2):191-6; discussion 196. PMID 16607899
- [Background] Baumgartner H, Falk V, Bax JJ, De Bonis M, Hamm C, Holm PJ, Iung B, Lancellotti P, Lansac E, Rodriguez Munoz D, Rosenhek R, Sjogren J, Tornos Mas P, Vahanian A, Walther T, Wendler O, Windecker S, Zamorano JL; ESC Scientific Document Group. 2017 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2017 Sep 21;38(36):2739-2791. doi: 10.1093/eurheartj/ehx391. No abstract available. PMID 28886619
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Fleisher LA, Jneid H, Mack MJ, McLeod CJ, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A. 2017 AHA/ACC Focused Update of the 2014 AHA/ACC Guideline for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2017 Jun 20;135(25):e1159-e1195. doi: 10.1161/CIR.0000000000000503. Epub 2017 Mar 15. No abstract available. PMID 28298458
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Williams M, Dewey T, Kapadia S, Babaliaros V, Thourani VH, Corso P, Pichard AD, Bavaria JE, Herrmann HC, Akin JJ, Anderson WN, Wang D, Pocock SJ; PARTNER Trial Investigators. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Engl J Med. 2011 Jun 9;364(23):2187-98. doi: 10.1056/NEJMoa1103510. Epub 2011 Jun 5. PMID 21639811
- [Background] Kapadia SR, Leon MB, Makkar RR, Tuzcu EM, Svensson LG, Kodali S, Webb JG, Mack MJ, Douglas PS, Thourani VH, Babaliaros VC, Herrmann HC, Szeto WY, Pichard AD, Williams MR, Fontana GP, Miller DC, Anderson WN, Akin JJ, Davidson MJ, Smith CR; PARTNER trial investigators. 5-year outcomes of transcatheter aortic valve replacement compared with standard treatment for patients with inoperable aortic stenosis (PARTNER 1): a randomised controlled trial. Lancet. 2015 Jun 20;385(9986):2485-91. doi: 10.1016/S0140-6736(15)60290-2. Epub 2015 Mar 15. PMID 25788231
- [Background] Popma JJ, Adams DH, Reardon MJ, Yakubov SJ, Kleiman NS, Heimansohn D, Hermiller J Jr, Hughes GC, Harrison JK, Coselli J, Diez J, Kafi A, Schreiber T, Gleason TG, Conte J, Buchbinder M, Deeb GM, Carabello B, Serruys PW, Chenoweth S, Oh JK; CoreValve United States Clinical Investigators. Transcatheter aortic valve replacement using a self-expanding bioprosthesis in patients with severe aortic stenosis at extreme risk for surgery. J Am Coll Cardiol. 2014 May 20;63(19):1972-81. doi: 10.1016/j.jacc.2014.02.556. Epub 2014 Mar 19. PMID 24657695
- [Background] Mack MJ, Leon MB, Smith CR, Miller DC, Moses JW, Tuzcu EM, Webb JG, Douglas PS, Anderson WN, Blackstone EH, Kodali SK, Makkar RR, Fontana GP, Kapadia S, Bavaria J, Hahn RT, Thourani VH, Babaliaros V, Pichard A, Herrmann HC, Brown DL, Williams M, Akin J, Davidson MJ, Svensson LG; PARTNER 1 trial investigators. 5-year outcomes of transcatheter aortic valve replacement or surgical aortic valve replacement for high surgical risk patients with aortic stenosis (PARTNER 1): a randomised controlled trial. Lancet. 2015 Jun 20;385(9986):2477-84. doi: 10.1016/S0140-6736(15)60308-7. Epub 2015 Mar 15. PMID 25788234
- [Background] Adams DH, Popma JJ, Reardon MJ, Yakubov SJ, Coselli JS, Deeb GM, Gleason TG, Buchbinder M, Hermiller J Jr, Kleiman NS, Chetcuti S, Heiser J, Merhi W, Zorn G, Tadros P, Robinson N, Petrossian G, Hughes GC, Harrison JK, Conte J, Maini B, Mumtaz M, Chenoweth S, Oh JK; U.S. CoreValve Clinical Investigators. Transcatheter aortic-valve replacement with a self-expanding prosthesis. N Engl J Med. 2014 May 8;370(19):1790-8. doi: 10.1056/NEJMoa1400590. Epub 2014 Mar 29. PMID 24678937
- [Background] Reardon MJ, Adams DH, Kleiman NS, Yakubov SJ, Coselli JS, Deeb GM, Gleason TG, Lee JS, Hermiller JB Jr, Chetcuti S, Heiser J, Merhi W, Zorn GL 3rd, Tadros P, Robinson N, Petrossian G, Hughes GC, Harrison JK, Maini B, Mumtaz M, Conte JV, Resar JR, Aharonian V, Pfeffer T, Oh JK, Qiao H, Popma JJ. 2-Year Outcomes in Patients Undergoing Surgical or Self-Expanding Transcatheter Aortic Valve Replacement. J Am Coll Cardiol. 2015 Jul 14;66(2):113-21. doi: 10.1016/j.jacc.2015.05.017. Epub 2015 Jun 5. PMID 26055947
- [Background] Latib A, Maisano F, Bertoldi L, Giacomini A, Shannon J, Cioni M, Ielasi A, Figini F, Tagaki K, Franco A, Covello RD, Grimaldi A, Spagnolo P, Buchannan GL, Carlino M, Chieffo A, Montorfano M, Alfieri O, Colombo A. Transcatheter vs surgical aortic valve replacement in intermediate-surgical-risk patients with aortic stenosis: a propensity score-matched case-control study. Am Heart J. 2012 Dec;164(6):910-7. doi: 10.1016/j.ahj.2012.09.005. Epub 2012 Oct 29. PMID 23194492
- [Background] Piazza N, Kalesan B, van Mieghem N, Head S, Wenaweser P, Carrel TP, Bleiziffer S, de Jaegere PP, Gahl B, Anderson RH, Kappetein AP, Lange R, Serruys PW, Windecker S, Juni P. A 3-center comparison of 1-year mortality outcomes between transcatheter aortic valve implantation and surgical aortic valve replacement on the basis of propensity score matching among intermediate-risk surgical patients. JACC Cardiovasc Interv. 2013 May;6(5):443-51. doi: 10.1016/j.jcin.2013.01.136. PMID 23702009
- [Background] D'Errigo P, Barbanti M, Ranucci M, Onorati F, Covello RD, Rosato S, Tamburino C, Santini F, Santoro G, Seccareccia F; OBSERVANT Research Group. Transcatheter aortic valve implantation versus surgical aortic valve replacement for severe aortic stenosis: results from an intermediate risk propensity-matched population of the Italian OBSERVANT study. Int J Cardiol. 2013 Sep 1;167(5):1945-52. doi: 10.1016/j.ijcard.2012.05.028. Epub 2012 May 26. PMID 22633667
- [Background] Leon MB, Smith CR, Mack MJ, Makkar RR, Svensson LG, Kodali SK, Thourani VH, Tuzcu EM, Miller DC, Herrmann HC, Doshi D, Cohen DJ, Pichard AD, Kapadia S, Dewey T, Babaliaros V, Szeto WY, Williams MR, Kereiakes D, Zajarias A, Greason KL, Whisenant BK, Hodson RW, Moses JW, Trento A, Brown DL, Fearon WF, Pibarot P, Hahn RT, Jaber WA, Anderson WN, Alu MC, Webb JG; PARTNER 2 Investigators. Transcatheter or Surgical Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med. 2016 Apr 28;374(17):1609-20. doi: 10.1056/NEJMoa1514616. Epub 2016 Apr 2. PMID 27040324
- [Background] Thourani VH, Kodali S, Makkar RR, Herrmann HC, Williams M, Babaliaros V, Smalling R, Lim S, Malaisrie SC, Kapadia S, Szeto WY, Greason KL, Kereiakes D, Ailawadi G, Whisenant BK, Devireddy C, Leipsic J, Hahn RT, Pibarot P, Weissman NJ, Jaber WA, Cohen DJ, Suri R, Tuzcu EM, Svensson LG, Webb JG, Moses JW, Mack MJ, Miller DC, Smith CR, Alu MC, Parvataneni R, D'Agostino RB Jr, Leon MB. Transcatheter aortic valve replacement versus surgical valve replacement in intermediate-risk patients: a propensity score analysis. Lancet. 2016 May 28;387(10034):2218-25. doi: 10.1016/S0140-6736(16)30073-3. Epub 2016 Apr 3. PMID 27053442
- [Background] Reardon MJ, Van Mieghem NM, Popma JJ, Kleiman NS, Sondergaard L, Mumtaz M, Adams DH, Deeb GM, Maini B, Gada H, Chetcuti S, Gleason T, Heiser J, Lange R, Merhi W, Oh JK, Olsen PS, Piazza N, Williams M, Windecker S, Yakubov SJ, Grube E, Makkar R, Lee JS, Conte J, Vang E, Nguyen H, Chang Y, Mugglin AS, Serruys PW, Kappetein AP; SURTAVI Investigators. Surgical or Transcatheter Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med. 2017 Apr 6;376(14):1321-1331. doi: 10.1056/NEJMoa1700456. Epub 2017 Mar 17. PMID 28304219
- [Background] Van Mieghem NM, Popma JJ, Deeb GM, Yakubov SJ, Serruys PW, Windecker S, Sondergaard L, Mumtaz M, Gada H, Chetcuti S, Kleiman NS, Kodali S, George I, Teefy P, Kiaii B, Oh JK, Kappetein AP, Chang Y, Mugglin AS, Reardon MJ; SURTAVI Trial Investigators. Complete 2-Year Results Confirm Bayesian Analysis of the SURTAVI Trial. JACC Cardiovasc Interv. 2020 Feb 10;13(3):323-331. doi: 10.1016/j.jcin.2019.10.043. PMID 32029248
- [Background] Mack MJ, Leon MB, Thourani VH, Makkar R, Kodali SK, Russo M, Kapadia SR, Malaisrie SC, Cohen DJ, Pibarot P, Leipsic J, Hahn RT, Blanke P, Williams MR, McCabe JM, Brown DL, Babaliaros V, Goldman S, Szeto WY, Genereux P, Pershad A, Pocock SJ, Alu MC, Webb JG, Smith CR; PARTNER 3 Investigators. Transcatheter Aortic-Valve Replacement with a Balloon-Expandable Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1695-1705. doi: 10.1056/NEJMoa1814052. Epub 2019 Mar 16. PMID 30883058
- [Background] Popma JJ, Deeb GM, Yakubov SJ, Mumtaz M, Gada H, O'Hair D, Bajwa T, Heiser JC, Merhi W, Kleiman NS, Askew J, Sorajja P, Rovin J, Chetcuti SJ, Adams DH, Teirstein PS, Zorn GL 3rd, Forrest JK, Tchetche D, Resar J, Walton A, Piazza N, Ramlawi B, Robinson N, Petrossian G, Gleason TG, Oh JK, Boulware MJ, Qiao H, Mugglin AS, Reardon MJ; Evolut Low Risk Trial Investigators. Transcatheter Aortic-Valve Replacement with a Self-Expanding Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1706-1715. doi: 10.1056/NEJMoa1816885. Epub 2019 Mar 16. PMID 30883053
- [Background] Chakos A, Wilson-Smith A, Arora S, Nguyen TC, Dhoble A, Tarantini G, Thielmann M, Vavalle JP, Wendt D, Yan TD, Tian DH. Long term outcomes of transcatheter aortic valve implantation (TAVI): a systematic review of 5-year survival and beyond. Ann Cardiothorac Surg. 2017 Sep;6(5):432-443. doi: 10.21037/acs.2017.09.10. PMID 29062738
- [Background] Horne A Jr, Reineck EA, Hasan RK, Resar JR, Chacko M. Transcatheter aortic valve replacement: historical perspectives, current evidence, and future directions. Am Heart J. 2014 Oct;168(4):414-23. doi: 10.1016/j.ahj.2014.07.017. Epub 2014 Jul 28. PMID 25262249
- [Background] Webb JG, Wood DA. Current status of transcatheter aortic valve replacement. J Am Coll Cardiol. 2012 Aug 7;60(6):483-92. doi: 10.1016/j.jacc.2012.01.071. Epub 2012 Jun 27. PMID 22749306
- [Background] Motloch LJ, Reda S, Rottlaender D, Khatib R, Muller-Ehmsen J, Seck C, Strauch J, Madershahian N, Erdmann E, Wahlers T, Hoppe UC. Postprocedural atrial fibrillation after transcatheter aortic valve implantation versus surgical aortic valve replacement. Ann Thorac Surg. 2012 Jan;93(1):124-31. doi: 10.1016/j.athoracsur.2011.08.078. Epub 2011 Nov 23. PMID 22115334
- [Background] Hahn RT, Pibarot P, Stewart WJ, Weissman NJ, Gopalakrishnan D, Keane MG, Anwaruddin S, Wang Z, Bilsker M, Lindman BR, Herrmann HC, Kodali SK, Makkar R, Thourani VH, Svensson LG, Akin JJ, Anderson WN, Leon MB, Douglas PS. Comparison of transcatheter and surgical aortic valve replacement in severe aortic stenosis: a longitudinal study of echocardiography parameters in cohort A of the PARTNER trial (placement of aortic transcatheter valves). J Am Coll Cardiol. 2013 Jun 25;61(25):2514-21. doi: 10.1016/j.jacc.2013.02.087. Epub 2013 Apr 23. PMID 23623915
- [Background] Pibarot P, Weissman NJ, Stewart WJ, Hahn RT, Lindman BR, McAndrew T, Kodali SK, Mack MJ, Thourani VH, Miller DC, Svensson LG, Herrmann HC, Smith CR, Rodes-Cabau J, Webb J, Lim S, Xu K, Hueter I, Douglas PS, Leon MB. Incidence and sequelae of prosthesis-patient mismatch in transcatheter versus surgical valve replacement in high-risk patients with severe aortic stenosis: a PARTNER trial cohort--a analysis. J Am Coll Cardiol. 2014 Sep 30;64(13):1323-34. doi: 10.1016/j.jacc.2014.06.1195. PMID 25257633
- [Background] Kodali S, Pibarot P, Douglas PS, Williams M, Xu K, Thourani V, Rihal CS, Zajarias A, Doshi D, Davidson M, Tuzcu EM, Stewart W, Weissman NJ, Svensson L, Greason K, Maniar H, Mack M, Anwaruddin S, Leon MB, Hahn RT. Paravalvular regurgitation after transcatheter aortic valve replacement with the Edwards sapien valve in the PARTNER trial: characterizing patients and impact on outcomes. Eur Heart J. 2015 Feb 14;36(7):449-56. doi: 10.1093/eurheartj/ehu384. Epub 2014 Oct 1. PMID 25273886
- [Background] Genereux P, Head SJ, Hahn R, Daneault B, Kodali S, Williams MR, van Mieghem NM, Alu MC, Serruys PW, Kappetein AP, Leon MB. Paravalvular leak after transcatheter aortic valve replacement: the new Achilles' heel? A comprehensive review of the literature. J Am Coll Cardiol. 2013 Mar 19;61(11):1125-36. doi: 10.1016/j.jacc.2012.08.1039. Epub 2013 Jan 30. PMID 23375925
- [Background] Manoharan G, Walton AS, Brecker SJ, Pasupati S, Blackman DJ, Qiao H, Meredith IT. Treatment of Symptomatic Severe Aortic Stenosis With a Novel Resheathable Supra-Annular Self-Expanding Transcatheter Aortic Valve System. JACC Cardiovasc Interv. 2015 Aug 24;8(10):1359-1367. doi: 10.1016/j.jcin.2015.05.015. PMID 26315740
- [Background] Husser O, Pellegrini C, Kessler T, Burgdorf C, Thaller H, Mayr NP, Ott I, Kasel AM, Schunkert H, Kastrati A, Hengstenberg C. Outcomes After Transcatheter Aortic Valve Replacement Using a Novel Balloon-Expandable Transcatheter Heart Valve: A Single-Center Experience. JACC Cardiovasc Interv. 2015 Dec 21;8(14):1809-16. doi: 10.1016/j.jcin.2015.08.014. PMID 26718512
- [Background] Binder RK, Stortecky S, Heg D, Tueller D, Jeger R, Toggweiler S, Pedrazzini G, Amann FW, Ferrari E, Noble S, Nietlispach F, Maisano F, Raber L, Roffi M, Grunenfelder J, Juni P, Huber C, Windecker S, Wenaweser P. Procedural Results and Clinical Outcomes of Transcatheter Aortic Valve Implantation in Switzerland: An Observational Cohort Study of Sapien 3 Versus Sapien XT Transcatheter Heart Valves. Circ Cardiovasc Interv. 2015 Oct;8(10):e002653. doi: 10.1161/CIRCINTERVENTIONS.115.002653. PMID 26453687
- [Background] Moretti C, D'Ascenzo F, Mennuni M, Taha S, Brambilla N, Nijhoff F, Fraccaro C, Barbanti M, Tamburino C, Tarantini G, Rossi ML, Presbitero P, Napodanno M, Stella P, Bedogni F, Omede P, Conrotto F, Montefusco A, Giordana F, Biondi Zoccai G, Agostoni P, D'Amico M, Rinaldi M, Marra S, Gaita F. Meta-analysis of comparison between self-expandable and balloon-expandable valves for patients having transcatheter aortic valve implantation. Am J Cardiol. 2015 Jun 15;115(12):1720-5. doi: 10.1016/j.amjcard.2015.03.015. Epub 2015 Mar 27. PMID 25890630
- [Background] Abdel-Wahab M, Mehilli J, Frerker C, Neumann FJ, Kurz T, Tolg R, Zachow D, Guerra E, Massberg S, Schafer U, El-Mawardy M, Richardt G; CHOICE investigators. Comparison of balloon-expandable vs self-expandable valves in patients undergoing transcatheter aortic valve replacement: the CHOICE randomized clinical trial. JAMA. 2014 Apr 16;311(15):1503-14. doi: 10.1001/jama.2014.3316. PMID 24682026
- [Background] Walther T, Hamm CW, Schuler G, Berkowitsch A, Kotting J, Mangner N, Mudra H, Beckmann A, Cremer J, Welz A, Lange R, Kuck KH, Mohr FW, Mollmann H; GARY Executive Board. Perioperative Results and Complications in 15,964 Transcatheter Aortic Valve Replacements: Prospective Data From the GARY Registry. J Am Coll Cardiol. 2015 May 26;65(20):2173-80. doi: 10.1016/j.jacc.2015.03.034. Epub 2015 Mar 15. PMID 25787198
- [Background] Mack MJ, Brennan JM, Brindis R, Carroll J, Edwards F, Grover F, Shahian D, Tuzcu EM, Peterson ED, Rumsfeld JS, Hewitt K, Shewan C, Michaels J, Christensen B, Christian A, O'Brien S, Holmes D; STS/ACC TVT Registry. Outcomes following transcatheter aortic valve replacement in the United States. JAMA. 2013 Nov 20;310(19):2069-77. doi: 10.1001/jama.2013.282043. PMID 24240934
- [Background] Athappan G, Gajulapalli RD, Sengodan P, Bhardwaj A, Ellis SG, Svensson L, Tuzcu EM, Kapadia SR. Influence of transcatheter aortic valve replacement strategy and valve design on stroke after transcatheter aortic valve replacement: a meta-analysis and systematic review of literature. J Am Coll Cardiol. 2014 May 27;63(20):2101-2110. doi: 10.1016/j.jacc.2014.02.540. Epub 2014 Mar 13. PMID 24632286
- [Background] Lansky AJ, Makkar R, Nazif T, Messe S, Forrest J, Sharma R, Schofer J, Linke A, Brown D, Dhoble A, Horwitz P, Zang M, DeMarco F, Rajagopal V, Dwyer MG, Zivadinov R, Stella P, Rovin J, Parise H, Kodali S, Baumbach A, Moses J. A randomized evaluation of the TriGuard HDH cerebral embolic protection device to Reduce the Impact of Cerebral Embolic LEsions after TransCatheter Aortic Valve ImplanTation: the REFLECT I trial. Eur Heart J. 2021 Jul 15;42(27):2670-2679. doi: 10.1093/eurheartj/ehab213. PMID 34000004
- [Background] Mollmann H, Hengstenberg C, Hilker M, Kerber S, Schafer U, Rudolph T, Linke A, Franz N, Kuntze T, Nef H, Kappert U, Walther T, Zembala MO, Toggweiler S, Kim WK. Real-world experience using the ACURATE neo prosthesis: 30-day outcomes of 1,000 patients enrolled in the SAVI TF registry. EuroIntervention. 2018 Feb 2;13(15):e1764-e1770. doi: 10.4244/EIJ-D-17-00628. PMID 29131801
- [Background] Kim WK, Mollmann H, Liebetrau C, Renker M, Rolf A, Simon P, Van Linden A, Arsalan M, Doss M, Hamm CW, Walther T. The ACURATE neo Transcatheter Heart Valve: A Comprehensive Analysis of Predictors of Procedural Outcome. JACC Cardiovasc Interv. 2018 Sep 10;11(17):1721-1729. doi: 10.1016/j.jcin.2018.04.039. Epub 2018 May 23. PMID 29803694
- [Background] Lanz J, Kim WK, Walther T, Burgdorf C, Mollmann H, Linke A, Redwood S, Thilo C, Hilker M, Joner M, Thiele H, Conzelmann L, Conradi L, Kerber S, Schymik G, Prendergast B, Husser O, Stortecky S, Heg D, Juni P, Windecker S, Pilgrim T; SCOPE I investigators. Safety and efficacy of a self-expanding versus a balloon-expandable bioprosthesis for transcatheter aortic valve replacement in patients with symptomatic severe aortic stenosis: a randomised non-inferiority trial. Lancet. 2019 Nov 2;394(10209):1619-1628. doi: 10.1016/S0140-6736(19)32220-2. Epub 2019 Sep 27. PMID 31570258
- [Background] ACURATE Neo AS study..
- [Background] Tamburino C, Bleiziffer S, Thiele H, Scholtz S, Hildick-Smith D, Cunnington M, Wolf A, Barbanti M, Tchetche D, Garot P, Pagnotta P, Gilard M, Bedogni F, Van Belle E, Vasa-Nicotera M, Chieffo A, Deutsch O, Kempfert J, Sondergaard L, Butter C, Trillo-Nouche R, Lotfi S, Mollmann H, Joner M, Abdel-Wahab M, Bogaerts K, Hengstenberg C, Capodanno D. Comparison of Self-Expanding Bioprostheses for Transcatheter Aortic Valve Replacement in Patients With Symptomatic Severe Aortic Stenosis: SCOPE 2 Randomized Clinical Trial. Circulation. 2020 Dec 22;142(25):2431-2442. doi: 10.1161/CIRCULATIONAHA.120.051547. Epub 2020 Oct 15. PMID 33054367
- [Background] Kim WK, Mollmann H, Liebetrau C, Renker M, Walther T, Hamm CW. Effectiveness and Safety of the ACURATE Neo Prosthesis in 1,000 Patients With Aortic Stenosis. Am J Cardiol. 2020 Sep 15;131:12-16. doi: 10.1016/j.amjcard.2020.05.044. Epub 2020 Jun 7. PMID 32622500
- [Background] Corcione N, Morello A, Ferraro P, Cimmino M, Testa L, Petronio AS, Iadanza A, Bartorelli AL, Berti S, Regazzoli D, Romagnoli E, Spaccarotella C, Tespili M, Pepe M, Frati G, Biondi-Zoccai G, Giordano A; Registro Italiano GISE sull'Impiantodi Valvola Aortica Percutanea (RISPEVA) Study Investigators. Comparing the Safety and Effectiveness of Five Leading New-Generation Devices for Transcatheter Aortic Valve Implantation: Twelve-Month Results From the RISPEVA Study. J Invasive Cardiol. 2021 May;33(5):E320-E329. doi: 10.25270/jic/20.00438. Epub 2021 Mar 19. PMID 33739300
- [Background] Costa et al. PCR LV 2018 Early clinical outcomes of three different second-generation transcatheter aortic valve prostheses
- [Background] Siqueira DA, Simonato M, Ramos AA, Bignoto T, Le Bihan D, Barreto RBM, Senra T, Pinto IM, Kambara AM, Santos MA, Viana R, Sousa AGMR, Abizaid AAC. Mid- to long-term clinical and echocardiographic outcomes after transcatheter aortic valve replacement with a new-generation, self-expandable system. Catheter Cardiovasc Interv. 2021 Jan 1;97(1):167-174. doi: 10.1002/ccd.28999. Epub 2020 May 23. PMID 32445607
- [Background] Ruck A. Results from the Early neo2 registry. ACURATE neo2 TAVI valve. EuroPCR 2021.
- [Background] VARC-3 WRITING COMMITTEE; Genereux P, Piazza N, Alu MC, Nazif T, Hahn RT, Pibarot P, Bax JJ, Leipsic JA, Blanke P, Blackstone EH, Finn MT, Kapadia S, Linke A, Mack MJ, Makkar R, Mehran R, Popma JJ, Reardon M, Rodes-Cabau J, Van Mieghem NM, Webb JG, Cohen DJ, Leon MB. Valve Academic Research Consortium 3: updated endpoint definitions for aortic valve clinical research. Eur Heart J. 2021 May 14;42(19):1825-1857. doi: 10.1093/eurheartj/ehaa799. PMID 33871579
- [Background] Brignole M, Auricchio A, Baron-Esquivias G, Bordachar P, Boriani G, Breithardt OA, Cleland J, Deharo JC, Delgado V, Elliott PM, Gorenek B, Israel CW, Leclercq C, Linde C, Mont L, Padeletti L, Sutton R, Vardas PE; ESC Committee for Practice Guidelines (CPG); Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Kirchhof P, Blomstrom-Lundqvist C, Badano LP, Aliyev F, Bansch D, Baumgartner H, Bsata W, Buser P, Charron P, Daubert JC, Dobreanu D, Faerestrand S, Hasdai D, Hoes AW, Le Heuzey JY, Mavrakis H, McDonagh T, Merino JL, Nawar MM, Nielsen JC, Pieske B, Poposka L, Ruschitzka F, Tendera M, Van Gelder IC, Wilson CM. 2013 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy: the Task Force on cardiac pacing and resynchronization therapy of the European Society of Cardiology (ESC). Developed in collaboration with the European Heart Rhythm Association (EHRA). Eur Heart J. 2013 Aug;34(29):2281-329. doi: 10.1093/eurheartj/eht150. Epub 2013 Jun 24. No abstract available. PMID 23801822
- [Background] SEC Working Group for the ESC 2015 Guidelines on the Management of Infective Endocarditis; Expert Reviewers for the ESC 2015 Guidelines on the Management of Infective Endocarditis; SEC Guidelines Committee. Comments on the ESC 2015 Guidelines for the Management of Infective Endocarditis. Rev Esp Cardiol (Engl Ed). 2016 Jan;69(1):7-10. doi: 10.1016/j.rec.2015.12.001. No abstract available. PMID 26748358
- [Background] Piepoli MF, Hoes AW, Agewall S, Albus C, Brotons C, Catapano AL, Cooney MT, Corra U, Cosyns B, Deaton C, Graham I, Hall MS, Hobbs FDR, Lochen ML, Lollgen H, Marques-Vidal P, Perk J, Prescott E, Redon J, Richter DJ, Sattar N, Smulders Y, Tiberi M, van der Worp HB, van Dis I, Verschuren WMM, Binno S; ESC Scientific Document Group. 2016 European Guidelines on cardiovascular disease prevention in clinical practice: The Sixth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of 10 societies and by invited experts)Developed with the special contribution of the European Association for Cardiovascular Prevention & Rehabilitation (EACPR). Eur Heart J. 2016 Aug 1;37(29):2315-2381. doi: 10.1093/eurheartj/ehw106. Epub 2016 May 23. No abstract available. PMID 27222591
- [Background] Stark, N.J., A new standard for medical device adverse event classification. J Clin Res Best Pract, 2009. 12: p. 1-8.
- [Background] Guidelines on medical devices, MEDDEV 2.7/3 - Clinical investigations: Serious adverse event reporting under directives 90/385/EEC and 93/42/EEC. European Commission. Directorate general for health and consumers. Consumer Affairs Cosmetics and Medical Devices. December 2010. http://ec.europa.eu/consumers/sectors/medical-devices/files/meddev/2_7_3_en.pdf.
- [Background] Ethical Principles for Medical Research Involving Human Subjects. WMA Declaration of Helsinki. Version October 2013. http://www.wma.net/en/30publications/10policies/b3/index.html.
- [Background] Guideline for good clinical practice E6(R1). International Conference on harmonisation of technical requirements for registration of pharmaceuticals for human use. June 10, 1996.
- [Background] Clinical investigation of medical devices for human subjects - Good clinical practice ISO 14155:2011. February 2011.
- [Background] Council directive 93/42/EEC concerning medical devices. The council of the european communities. June, 1993.
- [Background] Guidelines on medical devices, MEDDEV 2.7/4 - Guidelines on clinical investigation: A guide for manufacturers and notified bodies. . European Commission. Directorate general for health and consumers. Consumer Affairs Cosmetics and Medical Devices. December 2010. http://ec.europa.eu/consumers/sectors/medical-devices/files/meddev/2_7_4_en.pdf.